CLINICAL TRIAL: NCT03286179
Title: Standardizing Emergency Work-ups Around Risk Data (STEWARD): The CREST Network Chest Pain Project
Brief Title: Standardizing Emergency Work-ups Around Risk Data
Acronym: STEWARD
Status: Completed | Type: Observational
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: CN-16-2648
Record Dates: First submitted 2017-09-13; First posted 2017-09-18 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Acute Coronary Syndrome; Chest Pain; Risk Reduction
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: modified HEART score and/or Emergency Department Assessment of Chest pain Risk Score (EDACS) — Provision of estimated risk for major cardiac events at 60 days based on the modified HEART and/or EDACS, using KPNC specific estimates derived from an internal validation study

SUMMARY:
Chest pain is the second leading reason for emergency department (ED) visits in the United States. Resource utilization for this ED subpopulation is particularly high, in part due to a dearth of accepted standardized clinical approaches and general overestimation of risk on the part of both providers and patients. This prospective observational cohort study seeks to address this issue by providing externally validated risk scores for major adverse cardiac events using a web-based clinical decision support platform (RISTRA) embedded within the electronic health record at 13 Kaiser Permanente Northern California (KPNC) EDs over a 12-month period. The decision support will provide risk estimates specific to the KPNC patient population. This studies hypothesis is that the provision of more accurate risk estimation for major adverse cardiac events will improve informed decision making by both providers and patients, resulting in less provocative testing and lower ED lengths of stay amongst low risk patients, as well as improving medical management among non-low risk patients and decreasing future rates of major adverse cardiac events.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department chief complaint of chest pain or chest discomfort
* Clinical concern for possible cardiac ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to KPNC emergency departments with above elgibilty criteria
Sampling Method: Non-Probability Sample
Enrollment: 13419 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac event (MACE) | 12 months
  A composite outcome of either acute myocardial infarction, cardiac arrest, malignant arrhythmia, cardiac-related mortality

SECONDARY OUTCOMES:
Provocative and anatomic cardiac testing rates | 12 months
  Treadmill stress test, myocardial perfusion imaging, stress echocardiography, CT coronary angiography, catheter-based coronary angiography
Emergency department length of stay | 12 months
  Total hours spent in the emergency department among study eligible patients
Hospital admission rate | 12 months
  Percentage of hospital admissions among study eligible patients

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Kaiser Permanente Antioch Emergency Department, Antioch, California
  - Kaiser Permanente Fremont Emergency Department, Fremont, California
  - Kaiser Permanente Oakland Emergency Department, Oakland, California
  - Kaiser Permanente Richmond Emergency Department, Richmond, California
  - Kaiser Permanente Roseville Emergency Department, Roseville, California
  - Kaiser Permanente South Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente Sacramento Emergency Department, Sacramento, California
  - Kaiser Permanente San Francisco Emergency Department, San Francisco, California
  - Kaiser Permanente San Leandro Emergency Department, San Leandro, California
  - Kaiser Permanente San Rafael Emergency Department, San Rafael, California
  - Kaiser Permanente South San Francisco Emergency Department, South San Francisco, California
  - Kaiser Permanente Walnut Creek Emergency Department, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sabbatini AK, Nallamothu BK, Kocher KE. Reducing variation in hospital admissions from the emergency department for low-mortality conditions may produce savings. Health Aff (Millwood). 2014 Sep;33(9):1655-63. doi: 10.1377/hlthaff.2013.1318. PMID 25201672
- [Background] Venkatesh AK, Dai Y, Ross JS, Schuur JD, Capp R, Krumholz HM. Variation in US hospital emergency department admission rates by clinical condition. Med Care. 2015 Mar;53(3):237-44. doi: 10.1097/MLR.0000000000000261. PMID 25397965
- [Background] Newman DH, Ackerman B, Kraushar ML, Lederhandler MH, Masri A, Starikov A, Tsao DT, Meyers HP, Shah KH. Quantifying Patient-Physician Communication and Perceptions of Risk During Admissions for Possible Acute Coronary Syndromes. Ann Emerg Med. 2015 Jul;66(1):13-8, 18.e1. doi: 10.1016/j.annemergmed.2015.01.027. Epub 2015 Mar 4. PMID 25748480
- [Background] Than MP, Pickering JW, Aldous SJ, Cullen L, Frampton CM, Peacock WF, Jaffe AS, Goodacre SW, Richards AM, Ardagh MW, Deely JM, Florkowski CM, George P, Hamilton GJ, Jardine DL, Troughton RW, van Wyk P, Young JM, Bannister L, Lord SJ. Effectiveness of EDACS Versus ADAPT Accelerated Diagnostic Pathways for Chest Pain: A Pragmatic Randomized Controlled Trial Embedded Within Practice. Ann Emerg Med. 2016 Jul;68(1):93-102.e1. doi: 10.1016/j.annemergmed.2016.01.001. PMID 26947800
- [Background] Mahler SA, Riley RF, Hiestand BC, Russell GB, Hoekstra JW, Lefebvre CW, Nicks BA, Cline DM, Askew KL, Elliott SB, Herrington DM, Burke GL, Miller CD. The HEART Pathway randomized trial: identifying emergency department patients with acute chest pain for early discharge. Circ Cardiovasc Qual Outcomes. 2015 Mar;8(2):195-203. doi: 10.1161/CIRCOUTCOMES.114.001384. Epub 2015 Mar 3. PMID 25737484
- [Derived] Mark DG, Huang J, Ballard DW, Kene MV, Sax DR, Chettipally UK, Lin JS, Bouvet SC, Cotton DM, Anderson ML, McLachlan ID, Simon LE, Shan J, Rauchwerger AS, Vinson DR, Reed ME; Kaiser Permanente CREST Network Investigators [Link]. Graded Coronary Risk Stratification for Emergency Department Patients With Chest Pain: A Controlled Cohort Study. J Am Heart Assoc. 2021 Nov 16;10(22):e022539. doi: 10.1161/JAHA.121.022539. Epub 2021 Nov 6. PMID 34743565
- [Derived] Mark DG, Huang J, Kene MV, Sax DR, Cotton DM, Lin JS, Bouvet SC, Chettipally UK, Anderson ML, McLachlan ID, Simon LE, Shan J, Rauchwerger AS, Vinson DR, Ballard DW, Reed ME; Kaiser Permanente CREST Network Investigators. Prospective Validation and Comparative Analysis of Coronary Risk Stratification Strategies Among Emergency Department Patients With Chest Pain. J Am Heart Assoc. 2021 Apr 6;10(7):e020082. doi: 10.1161/JAHA.120.020082. Epub 2021 Mar 31. PMID 33787290